CLINICAL TRIAL: NCT02974387
Title: Randomized, Single Blinded Controlled Trial for Evaluation of the Safety and Efficacy of Loteprednol Versus Fluorometholone After Photorefractive Keratectomy for the Correction of Mild to Moderate Myopia, 3- Month Follow-up Study
Brief Title: Safety and Efficacy of Lotemax Versus FML in Subjects Undergoing PRK for the Correction of Mild to Moderate Myopia, 3- Month Follow-up Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr Salouti Eye Research Center (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SERCCT1
Record Dates: First submitted 2016-11-16; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Must be PRK Candidate
MeSH Terms: interventions — Fluorometholone; Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluorometholone(FMl) (Active Comparator): Patients will be randomized to the eye and will receive FML in one eye.
  Interventions: Drug: Fluorometholone(FML)
- Loteprednol (Lotemax) (Active Comparator): Patients will be randomized to the eye and will receive Lotemax in contralateral eye.
  Interventions: Drug: Loteprednol (Lotemax)

INTERVENTIONS:
Drug: Fluorometholone(FML)
  Arms: Fluorometholone(FMl)
Drug: Loteprednol (Lotemax)
  Arms: Loteprednol (Lotemax)

SUMMARY:
STUDY OBJECTIVE: To evaluate and compare the safety and efficacy of (corneal Wound Healing and Intraocular Pressure) Fluorometholone and Loteprednol after photorefractive keratectomy (PRK) surgery.

OVERALL STUDY DESIGN: Structure: Single-center, randomized, single blinded, contralateral (one eye receives FML, one eye Lotemax) Treatment Group: Patients will be randomized to the eye and will receive FML in one eye, Lotemax in contralateral eye Duration: 3 months Dosage/Dose Regimen: All patients will receive each one of the steroid agents 4 x a day for one month, 3 x a day for one month and 2 x a day for one month Study medication will be administered to the randomized eye through post op days according to mention protocol. Visit Schedule: baseline-screening, postop days 1, 7, 30 and then month 3th (through corneal re-epithelialization).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18-45 yrs of age, in good general health
* PRK candidate(Subjects willing and able to undergo bilateral PRK for the correction of their myopia. )
* Refractive error -1 to -8 diopters (spherical equivalent) at baseline
* Females of childbearing age must have a negative pregnancy test result at baseline. A female considered to be of non-childbearing potential is she is postmenopausal (no menses for 12 consecutive months) or is without a uterus.
* Ability to follow study instructions and likely to complete the entire course of the study(Subjects who are able to comply with all study procedures, including wearing a soft bandage contact lens in the immediate postoperative period. )
* Written informed consent will be obtained
* Written HIPPA authorization will be obtained
* Subjects with MRSE <6.0 D, with less than 2.0 D of astigmatism.
* Stable prescription in both eyes as defined by <0.25 D change over the preceding 2 years.

Exclusion Criteria:

* Uncontrolled systemic disease you mean if someone has controlled DM or rheumatic disease can be included
* Any active ocular disease, corneal abnormalities, lid abnormalities, or any ocular pathologies
* History of serious eye disease, trauma, or previous ocular surgery
* History of unstable myopia
* History of herpes keratitis
* Known allergy or hypersensitivity to the study medication
* Anticipated wearing of contact lenses in addition to the required bandage contact lens post-PRK. Patients who wear soft contact lenses should discontinue wearing them at least 7 days prior to baseline visit. Patients wearing RGP or hard contact lenses should discontinue wearing them at least 3 weeks prior to baseline visit.
* Females who are pregnant, breastfeeding, or trying to conceive.
* Keratoconus or keratoconus suspect
* Any condition or situation which, in the investigator's opinion, may put patient at significant risk or may confound the study results
* Subjects who have a past or present disease, which as judged by the investigator may affect the safety of the subject or the outcome of the study.
* Subjects who have previously had corneal surgery.
* Subjects with any ocular disease or corneal abnormality, including but not limited to:

  * Decreased corneal sensation / neurotrophic cornea;
  * Corneal vascularization;
  * Keratoconus;
  * Keratoconjunctivitis sicca requiring chronic treatment;
  * Lagophthalmos;
  * Blepharitis;
  * History of infectious keratitis;
  * History of glaucoma or intraocular pressure of >21 mmHg or use of glaucoma medications;
  * Significant dry eye disease that requires regular topical treatment;
  * Corneal thickness <480 µm at the thinnest point, and
  * Posterior elevation >40 micron.
  * Subjects who require any topical ophthalmic medication other than the pre- and postoperative regimen defined in the study protocol.
  * Subjects who are taking amiodarone, long acting anticholinergics, e.g., atropine, scopolamine, or medications or agents that can cause dry eye.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Time to re-epithelialization | 3-7 days
  Amount of days it takes for the cornea to re-epithelialize after PRK surgery, will be documented for each eye separately.

SECONDARY OUTCOMES:
Time to zero pain | 3-7 days
  Study subject will complete a questionnaire about their comfort levels at each postoperative visit, up to an including the 3-7 days post op exam.
Occurrence of enhancements | 3 months post operative
  Will document the number of requested/recommended enhancement procedures at the 3 month postoperative visit.
Incidence of adverse events | Day 1 up to day 90

IPD SHARING:
Plan to Share IPD: No